CLINICAL TRIAL: NCT06233396
Title: Uncertainty in Lung SBRT Simulation Based on 4DCT With Different Detector Widths
Brief Title: Feasibility Study of Radiation Therapy With Wide Detector 4DCT Scanning for Primary or Metastatic Lung Cancer
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc2022235
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-03

CONDITIONS: the Diffenence of Different Detector Row 4DCT，Especially in Artifects，Radiation Dose and Target Volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Extra 4DCT scan — Extra 4DCT scan after routine simulation

SUMMARY:
Currently there are very few studies using wide-body detectors for 4DCT to determine lung tumor volume and comparing them with conventional detector 4DCT images, and no prospective clinical trials comparing 4DCT images from different width detectors have been queried, therefore, in this study, we will prospectively explore in a body model and patients: 1) the degree of artifacts, tumor volume, and radiation dose of the 4DCT scans performed by different width detectors. differences, and scanning radiation dose. (ii) Whether there are differences in different tumor ITV outlining modalities on 4DCT with different detector widths.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in and sign the informed consent in person. 2. Over 18 years old, gender unlimited; 3. After imaging diagnosis of primary lung cancer or space-occupying lung lesions with oligometastases, MDT decided to treat SBRT 4. Clinical stage IA-IV (cT1-4N1-3M0-1); 5. No serious abnormality of blood system, heart, lung, liver, kidney function and immune deficiency; 6. Coagulation function: activated partial thromboplastin time (APTT) < the upper limit of normal 10 seconds, prothrombin time (PT) < the upper limit of normal 3 seconds, plasma fibrinogen 2-4g/L; 7. Hemoglobin ≥100g/L, WBC≥4×109/L, neutrophils ≥1.5×109/L, platelets ≥100×109/L 8. Bilirubin < 1.5 times the upper limit of normal value; Glutamic oxalic aminotransferase (ALT) & Glutamic pyruvic aminotransferase (AST) ≤1.5 times the upper limit of normal value; 9. Serum creatinine ≤1.5 times the upper limit of normal value; 10. The willingness of men or women of childbearing age to use contraception in the trial; 11. Physical condition score ECOG level 0 ~ 2; 12. Expected survival >3 months;

Exclusion Criteria:

* 1. Patients could not tolerate or were unwilling to undergo CT examination; 2. The primary lesion has undergone surgery or radiotherapy or chemotherapy or targeted or immunotherapy; 3. Subjects who have received other drug trials within the last 1 month; 4. People with severe allergic history or idiosyncrasies; 5. Patients with a history of severe lung or heart disease; 6. Severe comorbidities, such as uncontrolled hypertension, heart failure, etc.; 7. Pregnant or lactating women; 8. Previous history of malignant tumor; 9. Refusal or inability to sign informed consent to participate in the trial; 10. Currently or planning to participate in other clinical trials;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with primary or metastatic tumors in the lungs diagnosed by PETCT or puncture biopsy, in good general condition, who have completed gold standard implantation and are proposed to undergo SBRT
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
target volume | 2023.4-2024.1
  4DCT ITV delineation

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, National Clinical Research Center for Cancer, Key laboratory of Cancer Prevention and Therapy, Tianjin's Clinical Research Center for Cancer, Huan-Hu-Xi, Tianjin, Tianjin Municipality, China